CLINICAL TRIAL: NCT05969392
Title: Intradiscal Gelified Ethanol in Refractory Cervical Discogenic Pain : a Interventional, Prospective, Multi-center, Open-label Study.
Brief Title: Evaluation of Efficacy and Safety of Intradiscal Gelified Ethanol in Refractory Cervical Discogenic Pain
Acronym: DISCOCERV
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gelscom SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI01068
Record Dates: First submitted 2023-07-07; First posted 2023-08-01 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pain, Cervical; Discogenic Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intradiscal Gelified Ethanol Arm (Experimental): Patients who come with symptomatic cervical disc herniation or with cervical discogenic pain and meet the eligibility criteria.
  Interventions: Device: Intradiscal Gelified Ethanol (Discogel)

INTERVENTIONS:
Device: Intradiscal Gelified Ethanol (Discogel) — Intradiscal percutaneous injection of an intradiscal Gelified Ethanol

SUMMARY:
The purpose of this study is to assesse safety and efficacy of the Intradiscal Gelified Ethanol for treatment in refractory cervical discogenic pain.

DETAILED DESCRIPTION:
After being informed about the study and potential tisks, all patients giving written informed consent will undergo a inclusion visit (CT scan and X ray at least) for study entry. At Day 0, operation with Intradiscal Gelified Ethanol will be performed by the investigator. Follow visit will be performed at 3 months and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older;
* Pain refractory to conservative treatments for more than 2 months, non-surgical patients
* Cervicobrachialgia due to disc herniation
* Chronic discogenic pain (1 or 2 cervical discs) with concordant MRI;
* Patient agreeing to participate in the study and having given written consent;
* Patient enrolled in a health insurance plan.

Exclusion Criteria:

* Prior surgical treatment of the disc(s) studied;
* Sick leave of more than 12 months secondary to painful symptoms;
* Patient with Modic 1 score or more
* History of cognitive-behavioral disorders that could affect the completion of self-questionnaires;
* Local or systemic infection, or suspicion of infection;
* Severe coagulation disorders;
* Other inflammatory rheumatic disease;
* Severe underlying pathology with life expectancy <1 year;
* Women of childbearing age who are pregnant at the inclusion visit or who wish to become pregnant before the administration of the treatment (V0);
* Known allergy to contrast material and/or local anesthetic substances;
* Patients who cannot read or write Italian;
* Major person benefiting from a legal protection regime (guardianship, curatorship, safeguard of justice);

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
the mean change in pain intensity assessed by a verbal local rating scale (pain intensity numerical scale) between the pre-treatment measurement (inclusion visi) and the post-treatment measurement (Visit 2 at the 3 months) | 3 months
  In a 11-point numeric scale, 0 represents "NO PAIN" and 10 represents "EXTREME PAIN" (e.g., "pain as bad as you can imagine" and "worst pain imaginable").

SECONDARY OUTCOMES:
Change in pain cervical intensity using the verbal local rating scale [ | 12 months
  Scores range from 0-10. In a 11-point numeric scale, 0 represents "NO PAIN" and 10 represents "EXTREME PAIN" (e.g., "pain as bad as you can imagine" and "worst pain imaginable").
Change of consumption of painkillers | 12 months
  Number, frequency and dosage of pain relief treatments will be combine todescribe the difference in painkiller consumption before and after the operation
Incidence of complication and adverse event rates | 12 months
  Incidence of adverse event during 12 months after the treatment
Change in ability to manage everyday-life activity (Neck Disability Index (NDI) scale) [Time Frame : inclusion, 3 and 12 months after treatment]. | 12 months
  The Neck Disability Index (NDI) is used to measure pain-related disability associated with activities of daily living in people with neck pain (index between 0 and 50). The original report provided scoring intervals for interpretation, as follows: 0 - 4 = no disability, 5 - 14 = mild, 15 - 24 = moderate, 25 - 34 = severe, above 34 = complete. The NDI contains 10 items-7 related to activities of daily living, 2 related to pain, and 1 related to concentration.
Subjective evaluation MacNab | 12 months after treatment
  The MacNab's scale is layered into 4 levels (excellent, good, fair and poor) according to the patient's well-being after surgery or procedure.The scores were divided into the following four grades: 75-100% (excellent), 50-74% (good), 25-49% (fair) and 0-24% (poor). "Excellent" is defined as "No pain; no restriction of activity". "Good" is defined as "Occasional pain of sufficient severity to interfere with the patient's ability to do his normal work or his capacity to enjoy himself in leisure hours".

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Santissima Trinità Hospital Ascagliari, Cagliari
  - Azienda Ospedaliera Universitaria, Siena

IPD SHARING:
Plan to Share IPD: No
Confidential data (Pre-market Study trial)